CLINICAL TRIAL: NCT01750333
Title: Observational Retrospective Study on Correlation Between ET-1 and Ad in Obese Children
Brief Title: Study on Correlation Between Vascular ET-1 and Adiponectin in Pediatric Obesity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Monica Montagnani (Individual)
Responsible Party: Sponsor-Investigator, Monica Montagnani, Medical School Faculty Member - Professor of Pharmacology, Montagnani, Monica, M.D., Ph.D.
Organization: Montagnani, Monica, M.D., Ph.D. (Individual)
Other Study IDs: OBETAD-01
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: OBESITY; Endothelial Dysfunction; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — * serum
  * plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Lean children
- Overweight Children (OW)
- Obese children (Ob)

SUMMARY:
The aim of this study is to explore whether and how high circulating levels of endothelin-1 (ET-1) in obese and overweight children may contribute to impair adiponectin (Ad) production, release and vascular activity

ELIGIBILITY:
Inclusion Criteria:

* Children will be enrolled into lean, overweight or obese groups based on Body mass index (BMI) calculated according to standard methods. International standards for sex-and age-specific BMI centiles for subjects aged 2-18 years will be used. The 95th centile of BMI reference is the cut off point for childhood obesity. Overweight and obese children are defined as those with a BMI higher than the centile curves.

Exclusion Criteria:

* presence of renal, liver and/or cardiovascular diseases;
* hypertension;
* metabolic and/or endocrine disorders;
* genetic syndromes;
* histories of chronic allergies, acute infectious or inflammatory diseases during the last 3 months preceding the study

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: CHILDREN ATTENDING THE OUTPATIENT UNIT OF THE UNIVERSITY PEDIATRIC CLINIC
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Correlation between serum levels of ET-1 and Ad in lean, overweight and obese children | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Monica Montagnani, MD, PhD, Principal Investigator — University of Bari Medical School
Locations (1):
- University of Bari Medical School - Dept Biomedical Sciences and Human Oncology, Bari, Italy